CLINICAL TRIAL: NCT01033604
Title: Clinical Application of a Novel Dermal Substitute Based on Glycerol Preserved Allograft: GLYADERM
Brief Title: Glyaderm + Split Thickness Skin Graft Versus Split Thickness Skin Graft Alone in Full Thickness Skin Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Dutch Burnwound Foundation, Netherland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007/033
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Full Thickness Skin Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glyaderm and split skin graft (Experimental): Full thickness defects treated with Glyaderm and split skin graft.
  Interventions: Procedure: Glyaderm and split skin graft
- Split skin graft alone (Active Comparator): Full thickness defects treated with split skin graft alone.
  Interventions: Procedure: Split skin graft alone.

INTERVENTIONS:
Procedure: Glyaderm and split skin graft — Full thickness defects treated with Glyaderm and split skin graft.
  Arms: Glyaderm and split skin graft
Procedure: Split skin graft alone. — Full thickness defects treated with split skin graft alone.
  Arms: Split skin graft alone

SUMMARY:
The application of Glyaderm for skin restoration intends to provide a more stable wound closure with enhanced pliability and function of the skin and a more favourable scar. The dermal substitute would be affordable for widespread application in full thickness skin defects and burns.

Patients with burn wounds or large full thickness wounds will be evaluated before enrollment. All burn wounds that are not clearly full thickness on clinical assessment will be treated during the first 48 hours with a hydrocolloid paste and covered with a paraffin gauze dressing. This hydrocolloid paste combined with paraffin gauze will ensure maintenance of a moist wound environment for the first 48 hours prior to assessment by LDI and randomization. This is the standard treatment for all burns admitted to the Ghent Burn Centre.

Wounds will be photographed on a daily basis. In order to obtain an optimal preparation for LDI, the burn wounds will be meticulously debrided during dressing changes. LDI is most reliable between 48-72 hours. Patients whose burn wounds meet the inclusion criteria, i.e. full thickness burns with LDI values < 200 will be randomized to receive either GLYADERM and split skin graft versus split skin graft alone.

ELIGIBILITY:
Inclusion Criteria:

* All burn wounds with flux values measured by Laser Doppler Imaging, corresponding with an expected healing time longer than 28 days. Dark blue color on the palette of the LDI software with flux values below 200
* All clearly full thickness burns on clinical assessment done by two plastic surgeons and thereafter treated with Flammacerium®.
* Wounds treated with a hydrocolloid paste prior to LDI and with low flux values < 200
* All assessments are done during first days before final decision at day three
* Possibility to follow the complete treatment schedule until final graft take and subsequently wound healing and finally participation on complete follow-up schedule
* Informed consent has been obtained
* TBSA Full Thickness Burn < 40%

Exclusion Criteria:

* All burn wounds with flux values measured by Laser Doppler Imaging, corresponding with faster healing times ( flux values >200 )
* TBSA >40 %
* Not following the complete treatment schedule or missing some evaluations during the follow-up period
* Patient has any condition(s) that seriously compromises the patient's ability to complete this study.
* Patient has participated in another study utilizing an investigational drug within the previous 30 days
* Patient has one or more medical condition(s), diabetes, including renal, hepatic, hematologic, neurologic, or immune disease that in the opinion of the investigator would make the patient an inappropriate candidate for this study
* Patients wish to decline from the study
* No informed consent before start of the trial

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-09; Primary Completion 2012-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Comparison of healing time and percentage of autograft survival | After one week
Comparison in bacterial control in full thickness defects | On day 3,5 an 7 post application of Glyaderm
To assess the monitoring of dermal substitute ingrowth with Laser Doppler Imaging | On day 3, 5 and 7 post application of Glyaderm

SECONDARY OUTCOMES:
To evaluate the functional and cosmetic outcome of skin restoration of full thickness defects treated with Glyaderm and split skin graft versus split skin graft alone | 1 month, 3, 6 and 12 months post wound closure
Cost-effectiveness and Health related quality of life (i.e. cost utility analysis) | 1 month, 3, 6 and 12 months post wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Stan Monstrey, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] De Decker I, Hoeksema H, Verbelen J, De Coninck P, Speeckaert M, De Schepper S, Blondeel P, Pirayesh A, Monstrey S, Claes KEY. A single-stage bilayered skin reconstruction using Glyaderm(R) as an acellular dermal regeneration template results in improved scar quality: an intra-individual randomized controlled trial. Burns Trauma. 2023 May 2;11:tkad015. doi: 10.1093/burnst/tkad015. eCollection 2023. PMID 37143955
- See also: website of the University Hospital Ghent — http://www.uzgent.be